CLINICAL TRIAL: NCT05680948
Title: A Roll-Over Observational Study for the Extended Follow-Up of the Volunteers of the ISS T-003 Trial (ISS T-003 EF-UP2020)
Brief Title: Extended Follow-Up of the ISS T-003 Trial Volunteers (ISS T-003 EF-UP2020)
Acronym: T003EFUP2020
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Superiore di Sanità (Other)
Responsible Party: Sponsor
Other Study IDs: ISS T-003 EF-UP2020
Record Dates: First submitted 2022-12-05; First posted 2023-01-11 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
Keywords: HIV; HAART-treated participants; Tat protein; Therapeutic immunization
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled patients exiting the ISS T-003 EF-UP study: No intervention - No intervention is foreseen in this Observational Study

SUMMARY:
A further extension of the follow-up of the volunteers of the ISS T-003 trial is being conducted in order to evaluate the persistence of vaccine immunogenicity as well as of the immunological and virological effects induced by the therapeutic immunization with Tat after about 10 years from vaccination.

DETAILED DESCRIPTION:
The volunteers enrolled in the South African ISS T-003 trial (ClinicalTrials.gov NCT01513135; SANCTR: DOH-27-0211-3351) were recently enrolled in an observational study to extend the follow-up of the trial. The results of this study (ISS T-003 EF-UP, ClinicalTrials.gov NCT02712489; SANCTR: DOH-27-0615-4948) indicate the maintenance of anti-Tat Ab in a vast proposition of vaccinees.

The new roll-over observational study (ISS T-003 EF-UP2020; SANCTR: DOH-27-072022-7347) is to be conducted to further extend the follow-up of the participants of the ISS T-003 trial in order to evaluate the persistence of vaccine immunogenicity as well as of the immunological and virological effects induced by the therapeutic immunization with Tat after about 10 years from vaccination.

To this aim volunteers of the ISS T-003 study are included in a new 6-months study, with visits at weeks 0 and 24, during which the persistence and levels of anti-Tat antibodies (primary endpoint) and the CD4+ T-cell and HIV-1 plasma viraemia levels (secondary endpoint) will be evaluated. In addition, depending on the availability of residual specimens (PBMC, serum and plasma), further laboratory tests will be performed to investigate in-depth the immunological and virological profile of the volunteers. Clinical signs and symptoms of disease progression and AIDS-defining events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* previous participation in the ISS T-003 EF-UP study without withdrawal of consent;
* availability to participate in the ensuing extended follow-up study;
* signed informed consent.

Exclusion Criteria:

* The absence of any of the above criteria will exclude the participants from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Enrolment will be open to all patients who participated to the extended follow-up ("ISS T-003 EF-UP) of the therapeutic phase II trial of the Tat vaccine "ISS T-003".
  Potentially all patients enrolled in the ISS T-003 EF-UP study
Sampling Method: Non-Probability Sample
Enrollment: 179 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Anti-Tat humoral Immune responses | Week 0 and week 24
  Changes of anti-Tat serum antibody levels

SECONDARY OUTCOMES:
CD4+ T cells levels | Week 0 and week 24
  Evaluation of CD4+ T cell counts
HIV-1 plasma viremia | Week 0 and week 24
  Evaluation of HIV-1 RNA plasma levels
HIV-1 reservoir | Week 0 and week 24
  HIV-1 proviral DNA copies in blood

CONTACTS AND LOCATIONS:
Overall Officials: Maphoshane MN Nchabeleng, MD, Principal Investigator — Sefako Makgatho Health Sciences University - Mecru Clinical Research Unit (MeCRU),
Locations (1):
- Mecru Clinical Research Unit (MeCRU), Medunsa, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang HC, Samaniego F, Nair BC, Buonaguro L, Ensoli B. HIV-1 Tat protein exits from cells via a leaderless secretory pathway and binds to extracellular matrix-associated heparan sulfate proteoglycans through its basic region. AIDS. 1997 Oct;11(12):1421-31. doi: 10.1097/00002030-199712000-00006. PMID 9342064
- [Background] Fanales-Belasio E, Moretti S, Nappi F, Barillari G, Micheletti F, Cafaro A, Ensoli B. Native HIV-1 Tat protein targets monocyte-derived dendritic cells and enhances their maturation, function, and antigen-specific T cell responses. J Immunol. 2002 Jan 1;168(1):197-206. doi: 10.4049/jimmunol.168.1.197. PMID 11751963
- [Background] Rezza G, Fiorelli V, Dorrucci M, Ciccozzi M, Tripiciano A, Scoglio A, Collacchi B, Ruiz-Alvarez M, Giannetto C, Caputo A, Tomasoni L, Castelli F, Sciandra M, Sinicco A, Ensoli F, Butto S, Ensoli B. The presence of anti-Tat antibodies is predictive of long-term nonprogression to AIDS or severe immunodeficiency: findings in a cohort of HIV-1 seroconverters. J Infect Dis. 2005 Apr 15;191(8):1321-4. doi: 10.1086/428909. Epub 2005 Mar 14. PMID 15776379
- [Background] Re MC, Vignoli M, Furlini G, Gibellini D, Colangeli V, Vitone F, La Placa M. Antibodies against full-length Tat protein and some low-molecular-weight Tat-peptides correlate with low or undetectable viral load in HIV-1 seropositive patients. J Clin Virol. 2001 Apr;21(1):81-9. doi: 10.1016/s1386-6532(00)00189-x. PMID 11255101
- [Background] Reiss P, Lange JM, de Ronde A, de Wolf F, Dekker J, Debouck C, Goudsmit J. Speed of progression to AIDS and degree of antibody response to accessory gene products of HIV-1. J Med Virol. 1990 Mar;30(3):163-8. doi: 10.1002/jmv.1890300303. PMID 2341832
- [Background] Richardson MW, Mirchandani J, Duong J, Grimaldo S, Kocieda V, Hendel H, Khalili K, Zagury JF, Rappaport J. Antibodies to Tat and Vpr in the GRIV cohort: differential association with maintenance of long-term non-progression status in HIV-1 infection. Biomed Pharmacother. 2003 Jan;57(1):4-14. doi: 10.1016/s0753-3322(02)00327-x. PMID 12642031
- [Background] Cafaro A, Caputo A, Fracasso C, Maggiorella MT, Goletti D, Baroncelli S, Pace M, Sernicola L, Koanga-Mogtomo ML, Betti M, Borsetti A, Belli R, Akerblom L, Corrias F, Butto S, Heeney J, Verani P, Titti F, Ensoli B. Control of SHIV-89.6P-infection of cynomolgus monkeys by HIV-1 Tat protein vaccine. Nat Med. 1999 Jun;5(6):643-50. doi: 10.1038/9488. PMID 10371502
- [Background] Cafaro A, Bellino S, Titti F, Maggiorella MT, Sernicola L, Wiseman RW, Venzon D, Karl JA, O'Connor D, Monini P, Robert-Guroff M, Ensoli B. Impact of viral dose and major histocompatibility complex class IB haplotype on viral outcome in mauritian cynomolgus monkeys vaccinated with Tat upon challenge with simian/human immunodeficiency virus SHIV89.6P. J Virol. 2010 Sep;84(17):8953-8. doi: 10.1128/JVI.00377-10. Epub 2010 Jun 16. PMID 20554774
- [Background] Monini P, Cafaro A, Srivastava IK, Moretti S, Sharma VA, Andreini C, Chiozzini C, Ferrantelli F, Cossut MR, Tripiciano A, Nappi F, Longo O, Bellino S, Picconi O, Fanales-Belasio E, Borsetti A, Toschi E, Schiavoni I, Bacigalupo I, Kan E, Sernicola L, Maggiorella MT, Montin K, Porcu M, Leone P, Leone P, Collacchi B, Palladino C, Ridolfi B, Falchi M, Macchia I, Ulmer JB, Butto S, Sgadari C, Magnani M, Federico MP, Titti F, Banci L, Dallocchio F, Rappuoli R, Ensoli F, Barnett SW, Garaci E, Ensoli B. HIV-1 tat promotes integrin-mediated HIV transmission to dendritic cells by binding Env spikes and competes neutralization by anti-HIV antibodies. PLoS One. 2012;7(11):e48781. doi: 10.1371/journal.pone.0048781. Epub 2012 Nov 13. PMID 23152803
- [Background] Bellino S, Tripiciano A, Picconi O, Francavilla V, Longo O, Sgadari C, Paniccia G, Arancio A, Angarano G, Ladisa N, Lazzarin A, Tambussi G, Nozza S, Torti C, Foca E, Palamara G, Latini A, Sighinolfi L, Mazzotta F, Di Pietro M, Di Perri G, Bonora S, Mercurio VS, Mussini C, Gori A, Galli M, Monini P, Cafaro A, Ensoli F, Ensoli B. The presence of anti-Tat antibodies in HIV-infected individuals is associated with containment of CD4+ T-cell decay and viral load, and with delay of disease progression: results of a 3-year cohort study. Retrovirology. 2014 Jun 24;11:49. doi: 10.1186/1742-4690-11-49. PMID 24961156
- [Background] Cafaro A, Tripiciano A, Sgadari C, Bellino S, Picconi O, Longo O, Francavilla V, Butto S, Titti F, Monini P, Ensoli F, Ensoli B. Development of a novel AIDS vaccine: the HIV-1 transactivator of transcription protein vaccine. Expert Opin Biol Ther. 2015;15 Suppl 1:S13-29. doi: 10.1517/14712598.2015.1021328. Epub 2015 Jun 22. PMID 26096836
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Ensoli B, Cafaro A, Monini P, Marcotullio S, Ensoli F. Challenges in HIV Vaccine Research for Treatment and Prevention. Front Immunol. 2014 Sep 8;5:417. doi: 10.3389/fimmu.2014.00417. eCollection 2014. PMID 25250026
- [Background] Bellino S, Francavilla V, Longo O, Tripiciano A, Paniccia G, Arancio A, Fiorelli V, Scoglio A, Collacchi B, Campagna M, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Parallel conduction of the phase I preventive and therapeutic trials based on the Tat vaccine candidate. Rev Recent Clin Trials. 2009 Sep;4(3):195-204. doi: 10.2174/157488709789957529. PMID 20028332
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Monini P, Magnani M, Garaci E. The therapeutic phase I trial of the recombinant native HIV-1 Tat protein. AIDS. 2008 Oct 18;22(16):2207-9. doi: 10.1097/QAD.0b013e32831392d4. PMID 18832884
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Tripiciano A, Longo O, Bellino S, Francavilla V, Paniccia G, Arancio A, Scoglio A, Collacchi B, Ruiz Alvarez MJ, Tambussi G, Tassan Din C, Palamara G, Latini A, Antinori A, D'Offizi G, Giuliani M, Giulianelli M, Carta M, Monini P, Magnani M, Garaci E. The preventive phase I trial with the HIV-1 Tat-based vaccine. Vaccine. 2009 Dec 11;28(2):371-8. doi: 10.1016/j.vaccine.2009.10.038. Epub 2009 Oct 29. PMID 19879233
- [Background] Longo O, Tripiciano A, Fiorelli V, Bellino S, Scoglio A, Collacchi B, Alvarez MJ, Francavilla V, Arancio A, Paniccia G, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Phase I therapeutic trial of the HIV-1 Tat protein and long term follow-up. Vaccine. 2009 May 26;27(25-26):3306-12. doi: 10.1016/j.vaccine.2009.01.090. Epub 2009 Feb 7. PMID 19208456
- [Background] Ensoli B, Bellino S, Tripiciano A, Longo O, Francavilla V, Marcotullio S, Cafaro A, Picconi O, Paniccia G, Scoglio A, Arancio A, Ariola C, Ruiz Alvarez MJ, Campagna M, Scaramuzzi D, Iori C, Esposito R, Mussini C, Ghinelli F, Sighinolfi L, Palamara G, Latini A, Angarano G, Ladisa N, Soscia F, Mercurio VS, Lazzarin A, Tambussi G, Visintini R, Mazzotta F, Di Pietro M, Galli M, Rusconi S, Carosi G, Torti C, Di Perri G, Bonora S, Ensoli F, Garaci E. Therapeutic immunization with HIV-1 Tat reduces immune activation and loss of regulatory T-cells and improves immune function in subjects on HAART. PLoS One. 2010 Nov 11;5(11):e13540. doi: 10.1371/journal.pone.0013540. PMID 21085635
- [Background] Ensoli F, Cafaro A, Casabianca A, Tripiciano A, Bellino S, Longo O, Francavilla V, Picconi O, Sgadari C, Moretti S, Cossut MR, Arancio A, Orlandi C, Sernicola L, Maggiorella MT, Paniccia G, Mussini C, Lazzarin A, Sighinolfi L, Palamara G, Gori A, Angarano G, Di Pietro M, Galli M, Mercurio VS, Castelli F, Di Perri G, Monini P, Magnani M, Garaci E, Ensoli B. HIV-1 Tat immunization restores immune homeostasis and attacks the HAART-resistant blood HIV DNA: results of a randomized phase II exploratory clinical trial. Retrovirology. 2015 Apr 29;12:33. doi: 10.1186/s12977-015-0151-y. PMID 25924841
- [Background] Sgadari C, Monini P, Tripiciano A, Picconi O, Casabianca A, Orlandi C, Moretti S, Francavilla V, Arancio A, Paniccia G, Campagna M, Bellino S, Meschiari M, Nozza S, Sighinolfi L, Latini A, Muscatello A, Saracino A, Di Pietro M, Galli M, Cafaro A, Magnani M, Ensoli F, Ensoli B. Continued Decay of HIV Proviral DNA Upon Vaccination With HIV-1 Tat of Subjects on Long-Term ART: An 8-Year Follow-Up Study. Front Immunol. 2019 Feb 13;10:233. doi: 10.3389/fimmu.2019.00233. eCollection 2019. PMID 30815001
- [Result] Ensoli B, Nchabeleng M, Ensoli F, Tripiciano A, Bellino S, Picconi O, Sgadari C, Longo O, Tavoschi L, Joffe D, Cafaro A, Francavilla V, Moretti S, Pavone Cossut MR, Collacchi B, Arancio A, Paniccia G, Casabianca A, Magnani M, Butto S, Levendal E, Ndimande JV, Asia B, Pillay Y, Garaci E, Monini P; SMU-MeCRU study group. HIV-Tat immunization induces cross-clade neutralizing antibodies and CD4(+) T cell increases in antiretroviral-treated South African volunteers: a randomized phase II clinical trial. Retrovirology. 2016 Jun 9;13(1):34. doi: 10.1186/s12977-016-0261-1. PMID 27277839
- See also: ISS CNAIDS Website — https://www.iss.it/web/guest/centro-nazionale-per-la-ricerca-su-hiv/aids